CLINICAL TRIAL: NCT02562131
Title: 18F-Fluciclovine PET/MRI for Detection of Recurrent Prostate Cancer After Radical Treatment
Brief Title: PET-MR-PSA Prostate Cancer Recidive Study
Acronym: PET-MR-PSA
Status: Active, not recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/163-4
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer Recurrent
Keywords: PET-MR; recidive; PET/MR imaging; 18F-Fluciclovine; radical treatment; recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Simultaneous PET/MRI has the potential to improve the detection accuracy in recurrent prostate cancer, since it combines the excellent soft-tissue contrast of MRI with the high molecular sensitivity of PET in a single imaging session. The aim of this study is to evaluate the sensitivity and specificity of simultaneous 18F-Fluciclovine PET/MRI for detection of recurrent prostate cancer.

DETAILED DESCRIPTION:
The patients follow standard treatment and follow-up after the PET/MRI exam, which will be determined by the patient's treating urologist and/or oncologist. Data from histopathology, clinical follow-up and follow-up imaging will be collected to establish a reference standard that defines the presence or absence of disease for each patient. The imaging findings will be compared with the reference standard to assess the sensitivity and specificity. The diagnostic accuracy of combined PET/MRI and MRI-only (the current clinical standard) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* the criteria for biochemical relapse in accordance with the European Association of Urology (EAU) guidelines on prostate cancer must be fulfilled (two consecutive measurements with PSA > 0.2 ng/ml following radical prostatectomy or PSA > 2.0 ng/ml above the nadir following definitive radiotherapy)
* potential candidates for salvage treatment based on age and co-morbidity.

Exclusion Criteria:

* general contra-indications for a PET/MRI exam (pacemaker, aneurysm clips, any form of metal in the body, or severe claustrophobia)
* impaired renal function defined as estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim in 2 years is 80 prostate cancer patients with biochemical relapse following radical treatment, or patients with persistently elevated PSA levels after radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Detection of recurrent prostate cancer by simultaneous 18F-Fluciclovine PET/MRI. | 10 years
  Relevant patient information will be collected until 2027, 10 years after the last PET/MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Tone F Bathen, PhD, Principal Investigator — The Norwegian University of Science and Technology (NTNU)
Locations (1):
- St Olavs Hospital, PET center, Trondheim, Norway